CLINICAL TRIAL: NCT05559866
Title: Hybrid Argon Plasma Coagulation and Endoscopic Sleeve Gastroplasty Trial (HAPCET): A Single-center Randomized Controlled Trial
Brief Title: Hybrid Argon Plasma Coagulation and Endoscopic Sleeve Gastroplasty Trial
Acronym: HAPCET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Erbe Elektromedizin GmbH (Industry)
Responsible Party: Principal Investigator, Omar Ghanem, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-001202
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Obesity
Keywords: ESG; Hybrid APC
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Group: ESG (Active Comparator): Subjects will undergo ESG utilizing approved device alone
  Interventions: Device: Apollo ESG
- Treatment Group: ESG + HAPC (Experimental): Subjects will undergo ESG as approved and on-label while also utilizing Hybrid APC approved and on-label.
  Interventions: Device: Apollo ESG with ERBE HAPC

INTERVENTIONS:
Device: Apollo ESG with ERBE HAPC — Utilizing two approved devices in combination to assess durability of suturing.
  Arms: Treatment Group: ESG + HAPC
Device: Apollo ESG — Using only Apollo ESG as approved per label.
  Arms: Control Group: ESG

SUMMARY:
This study is being done to evaluate the safety and effectiveness of combined Hybrid Argon Plasma Coagulation (HAPC) and Endoscopic Sleeve Gastroplasty (ESG) for weight loss and improvement in obesity-related co-morbidities compared to ESG alone in participants with a BMI ≥ 30 and ≤40 kg/m² who have failed to achieve and maintain weight loss with a non-surgical program.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 and ≤40 kg/m²
* Willingness to comply with the substantial lifelong dietary restrictions required by the procedure.
* History of failure with non-surgical weight-loss methods.
* Willingness to follow protocol requirements, including signed informed consent, routine follow-up schedule, completing laboratory tests, and completing diet counseling.
* Residing within a reasonable distance from the investigator's office and able to travel to the investigator to complete all routine follow-up visits.
* Ability to give informed consent.
* Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods.

Exclusion Criteria:

* History of foregut or gastrointestinal (GI) surgery (except uncomplicated cholecystectomy or appendectomy).
* Prior gastrointestinal surgery with sequelae, i.e. obstruction, and/or adhesive peritonitis or known abdominal adhesions.
* Prior open or laparoscopic bariatric surgery.
* Prior surgery of any kind on the esophagus, stomach, or any type of hiatal hernia surgery.
* Any inflammatory disease of the gastrointestinal tract including severe (LA Grade C or D) esophagitis, Barrett's esophagus, gastric ulceration, duodenal ulceration, cancer, or specific inflammatory disease such as Crohn's disease or celiac disease.
* Potential upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the gastrointestinal tract such as atresias or stenoses.
* Gastrointestinal stromal tumors, history of premalignant gastric lesions (intestinal metaplasia), history of familial and nan-familial adenomatous syndromes.
* A gastric mass or gastric polyps > 1 cm in size.
* A hiatal hernia > 4cm of axial displacement of the z-line above the diaphragm or severe or intractable gastro-esophageal reflux symptoms.
* A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the endoscope.
* Achalasia or any other severe esophageal motility disorder
* Severe coagulopathy.
* Insulin-dependent diabetes (either Type 1 or Type 2) or a significant likelihood of requiring insulin treatment in the following 12 months or a HgbA1C≥9.
* Subjects with any serious health condition unrelated to their weight that would increase the risk of endoscopy.
* Chronic abdominal pain.
* Motility disorders of the GI tract such as gross esophageal motility disorders, gastroparesis or intractable constipation.
* Hepatic insufficiency or cirrhosis.
* Use of an intragastric device prior to this study due to the increased thickness of the stomach wall preventing effective suturing.
* Active psychological issues preventing participation in a life-style modification program as determined by a psychologist.
* Patients unwilling to participate in an established medically supervised diet and behavior modification program, with routine medical follow-up.
* Patients receiving daily prescribed treatment with high dose aspirin (> 81mg daily), anti-inflammatory agents, anticoagulants, or other gastric irritants.
* Patients who are unable or unwilling to take prescribed proton pump inhibitor medication.
* Patients who are pregnant or breast-feeding.
* Patients currently taking weight-loss medications or other therapies for weight loss within the prior 6 months.
* Subjects with severe cardiopulmonary disease or other serious organic disease which might include known history of coronary artery disease, myocardial infarction within the past 6 months, poorly controlled hypertension, required use of NSAIDs.
* Subjects taking medications on specified hourly intervals that may be affected by changes to gastric emptying, such as anti-seizure or anti-arrhythmic medications.
* Subjects who are taking corticosteroids, immunosuppressants, and narcotics.
* Symptomatic congestive heart failure, cardiac arrhythmia, or unstable coronary artery disease.
* Pre-existing respiratory disease such as moderate or severe chronic obstructive pulmonary disease (COPD) requiring steroids, pneumonia, or cancer.
* Diagnosis of autoimmune connective tissue disorder (e.g. Systemic lupus erythematosus, scleroderma) or immunocompromised.
* Specific diagnosed genetic disorder such as Prader Willi syndrome.
* Eating disorders including night eating syndrome (NES), bulimia, binge eating disorder, or compulsive overeating.
* Known history of endocrine disorders affecting weight such as uncontrolled hypothyroidism.
* At the discretion of the PI for subject safety
* If minority inclusion population target of 10% has not been reached by the 90% enrollment mark (example 21 of 24 subjects), the remaining enrollments will be reserved for minority subjects (example 3 of 24 subjects).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2025-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Ghanem, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at a single center, Mayo Clinic Rochester. Recruitment was primarily achieved through direct advertising leading subjects to self-refer, as well as physician referrals. 45 patients were enrolled, 24 were randomized and underwent study treatment either in the ESG arm or the ESG-HAPC arm. The last patient was enrolled in November of 2023 and the last treatment procedure was completed in January of 2024.
Pre-assignment Details: Of the 45 enrolled participants only 24 moved forward to randomization and treatment. Reasons for exclusion included non-qualifying BMI, disqualifying psychological intake findings, findings on laboratory testing or MRI, and patient refusal to complete screening activities.
Period: Overall Study
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Started | 12 | 12
6 Month Post-procedure Visit | 12 | 12
12 Month Post-procedure Visit | 11 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (6.2) | 47.8 (9.2) | 45.5 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 12 | 12 | 24
BMI [Mean (Standard Deviation); unit: kg/m²] — Body Mass Index
  kg/m² | 36.6 (2.4) | 36.6 (2.1) | 36.6 (2.22)
Hypertension [Count of Participants; unit: Participants] — Comorbidity
  Participants | 0 | 3 | 3
Hyperlipidemia [Count of Participants; unit: Participants] — Comorbidity
  Participants | 3 | 3 | 6
Sleep Apnea [Count of Participants; unit: Participants] — Comorbidity
  Participants | 0 | 2 | 2
Mood Disorder [Count of Participants; unit: Participants] | 6 | 5 | 11
Current smoker [Count of Participants; unit: Participants] | 0 | 0 | 0
Current alcohol use [Count of Participants; unit: Participants] | 10 | 6 | 16
Type 2 diabetes mellitus [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Durability
Description: The primary outcomes are durability of plications and endoscopic sutures on repeat endoscopy at 6 months, in the two randomized arms.
  Endoscopic scale runs from 0 to 3. A lower score indicates less durability and a higher score indicates greater durability.
Time Frame: 6 months
Population: One participant in the ESG arm elected not to undergo the endoscopy at which the durability assessment is performed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Number analyzed (Participants) | 11 | 12
Score on a scale
  Proximal Stomach - Tubular form | 1.2 (0.1) | 3.0 (0.12)
  Proximal stomach - Bridging fibrosis | 1.4 (0.7) | 3.0 (0.0)
  Proximal stomach - accommodation to insufflation | 1.4 (0.7) | 3.0 (0)
  Mid-stomach - tubular form | 2.8 (0.4) | 1.8 (0.7)
  Mid Stomach - bridging fibrosis | 2.8 (0.4) | 1.9 (0.7)
  Mid Stomach - accommodation to insufflation | 2.8 (0.4) | 1.8 (0.6)
  Distal Stomach - tubular form | 1.3 (0.6) | 2.2 (0.6)
  Distal stomach - bridging fibrosis | 1.5 (0.7) | 2.0 (0.7)
  Distal stomach - accommodation to insufflation | 1.2 (0.4) | 1.9 (0.5)
Statistical Analysis 1: Comparison: Control Group: ESG vs Treatment Group: ESG + HAPC; Scores from the proximal stomach, mid-stomach and distal stomach in the control and treatment groups were analyzed to determine if there was a significant difference between the mean difference in durability scores for the control and treatment groups; Test type: Other — Variance; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [.31 to .74]

2. Secondary Outcome: Percent Total Body Weight Loss (%TBWL)
Description: Compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis. Percent total body weight loss was analyzed for variance between treatment and control groups accounting for gender and starting obesity class (determined by starting body mass index).
  Total body weight loss is calculated as follows: Total Body Weight Loss (%) = [ (Starting Weight - Current Weight) / Starting Weight ] × 100
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Number analyzed (Participants) | 12 | 12
Percentage | 19.5 (6.2) | 18.8 (4.4)
Statistical Analysis 1: Comparison: Control Group: ESG vs Treatment Group: ESG + HAPC; Test type: Other — Variance; p = 1.00, ANCOVA; Mean Difference (Final Values) = 19.125, 95% CI 2-sided [19.125 to 19.125], Standard Error of Mean 0.00000130

3. Secondary Outcome: Percent Excess Weight Loss (%EWL)
Description: Compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis. Percent excess weight loss was analyzed for variance between treatment and control groups accounting for gender and starting obesity class (determined by starting body mass index).
  % EWL = (actual weight lost / excess body weight) x 100 Where excess body weight represents the difference in starting weight and ideal weight (weight corresponding to a body mass index of 25 kg/m^2)
Time Frame: 6 and 12 month
Population: All 24 patients completed their weigh in at 6 months, 2 patients in the ESG arm did not weigh in at 12 months (one due to patient withdrawal, one due to patient noncompliance).
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Number analyzed (Participants) | 12 | 12
Percentage
  6 Months | 101.5 (73.68) | 88.69 (70.92)
  12 Months: number analyzed (Participants) | 10 | 12
  12 Months | 125.49 (87.96) | 187.15 (200.95)
Statistical Analysis 1: Comparison: Control Group: ESG vs Treatment Group: ESG + HAPC; Test type: Other — Variance; p = 0.757, ANCOVA — alpha = 0.05; 1 degree of freedom

4. Secondary Outcome: Blood Pressure
Description: Compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis. Blood pressure scores analyzed for variance between treatment and control groups accounting for gender and starting obesity class (determined by starting body mass index).
Time Frame: 6 month
Measure: Mean (Full Range); unit: mm HG
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Number analyzed (Participants) | 12 | 12
mm HG
  Systolic | 113.8 [101 to 125] | 119.8 [99 to 150]
  Diastolic | 73.9 [57 to 85] | 76.3 [63 to 99]
Statistical Analysis 1: Comparison: Control Group: ESG vs Treatment Group: ESG + HAPC; Test type: Other — Variance; p = 0.271, ANCOVA — Alpha = 0.05; 1 degree of freedom

5. Secondary Outcome: Percentage of Glycated Hemoglobin (% HbA1c)
Description: Compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Number analyzed (Participants) | 12 | 12
Percentage | 4.9 (0.28) | 5.1 (0.22)
Statistical Analysis 1: Comparison: Control Group: ESG vs Treatment Group: ESG + HAPC; Test type: Other — Variance; p = 0.29, ANCOVA — alpha = 0.05; 1 degree of freedom

6. Secondary Outcome: Questionnaire: Short Form (36) Health Survey [SF-36]
Description: Compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis.
  8 quality of life domains assessed, domains scores range 0-100 with a lower score indicating a worse outcome, and a higher score indicating a better outcome.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Number analyzed (Participants) | 12 | 12
Score on a scale
  Physical Functioning | 98.3 (3.3) | 89.6 (14.5)
  Role Limitations Due to Physical Health | 97.9 (7.2) | 93.8 (21.7)
  Bodily Pain | 87.7 (16.6) | 80.6 (22.7)
  General Health Perceptions | 77.5 (13.1) | 79.2 (7.9)
  Vitality (Energy and Fatigue) | 60.4 (19.1) | 75.4 (13.2)
  Social Functioning | 89.6 (19.1) | 89.6 (17.5)
  Role Limitations Due to Emotional Problems | 88.88 (29.6) | 100 (0)
  Emotional well-being | 81.7 (15.8) | 86.7 (13.2)
Statistical Analysis 1: Comparison: Control Group: ESG vs Treatment Group: ESG + HAPC; Test type: Other — Variance; p = 0.72, ANCOVA — alpha = 0.05; 1 degree of freedom

7. Secondary Outcome: Questionnaire: Impact of Weight on Quality of Life (IWQOL)
Description: Compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis.
  5 quality of life domains are scored, a higher score indicates higher quality of life relative to that domain and lower score indicates worse quality of life relative to that domain.
  Physical function domain (11 items scored 1-5) total scores ranging 11-55 Self-esteem domain (seven items scored 1-5) total scores ranging 7-35 Sexual life domain (four items each scored 1-5) total scores ranging 4-20 Public distress domain (five items each scored 1-5) total scores ranging 5-25 Work-related domain (four items each scored 1-5) total scores ranging 4-20
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Number analyzed (Participants) | 12 | 12
Score on a scale
  Physical function score | 13.08 (3.6) | 12.91 (2.5)
  Self-esteem score | 14 (4.8) | 12 (6.3)
  Sexual life score | 7.3 (3.0) | 6.6 (3.1)
  Public distress score | 5.4 (1.5) | 5.25 (0.6)
  Work-related score | 4 (0.7) | 4.08 (0.3)
Statistical Analysis 1: Comparison: Control Group: ESG vs Treatment Group: ESG + HAPC; Test type: Other — Variance; p = 0.41, ANCOVA — alpha = 0.05; 1 degree of freedom

8. Secondary Outcome: Questionnaire: Patient Health Questionnaire-9 (PHQ-9)
Description: Compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis.
  Score range 0-27, with a higher score indicating more severe symptoms and a lower score indicating less severe or no symptoms.
Time Frame: 6 month
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Number analyzed (Participants) | 12 | 12
Score on a scale | 1.8 [0 to 5] | 1.1 [0 to 6]
Statistical Analysis 1: Comparison: Control Group: ESG vs Treatment Group: ESG + HAPC; Test type: Other — Variance; p = 0.53, ANCOVA — alpha = 0.05; 1 degree of freedom

9. Secondary Outcome: Questionnaire: Eating Behavior
Description: Compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis.
  Scored across three behavioral domains, higher scores in each subscale indicate a greater tendency towards that particular eating behavior.
  Cognitive Restraint Score range 6-28 Uncontrolled Eating Score range 9-36 Emotional Eating Score range 3-12
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Number analyzed (Participants) | 12 | 12
Score on a scale
  Cognitive restraint score | 18.4 (2.4) | 18.8 (3.0)
  Uncontrolled eating score | 14.1 (4.1) | 11.6 (3.1)
  Emotional eating score | 5.3 (2.3) | 4.2 (1.3)
Statistical Analysis 1: Comparison: Control Group: ESG vs Treatment Group: ESG + HAPC; Test type: Other — Variance; p = 0.91, ANCOVA — alpha = 0.05; 1 degree of freedom

10. Secondary Outcome: Binary Outcome: ≥25% Reduction in Percent Excess Weight Loss (%EWL)
Description: Compared between treatment arms by Pearson Chi-square test.
  % EWL = (actual weight lost / excess body weight) x 100 Where excess body weight represents the difference in starting weight and ideal weight (weight corresponding to a body mass index of 25 kg/m^2)
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Number analyzed (Participants) | 12 | 12
Participants | 11 | 12
Statistical Analysis 1: Comparison: Control Group: ESG vs Treatment Group: ESG + HAPC; Test type: Other; p = 0.307, Chi-squared; Chi-Square: 1.043478

11. Secondary Outcome: Binary Outcome: Incidence of Esophagitis
Description: Compared between treatment arms by Pearson Chi-square test.
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
Number analyzed (Participants) | 11 | 12
Participants | 0 | 0
Statistical Analysis 1: Comparison: Control Group: ESG vs Treatment Group: ESG + HAPC; Test type: Other — Association; Unable to perform Chi-Square test as data in both categorical sets was identical - there is no variation to test

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow up, up to 52 weeks post-treatment
Arm/Group | Control Group: ESG | Treatment Group: ESG + HAPC
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group: ESG (N=12) | Treatment Group: ESG + HAPC (N=12)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (4)
GERD (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Patchy tongue lesions (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a pilot trial and therefore no formal power analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT05559866/Prot_SAP_000.pdf